CLINICAL TRIAL: NCT02095886
Title: Assessment of BMS-955176 Bioavailability From a Micronized Crystalline Tablet Relative to a Spray-Dried Dispersion Suspension and Assessment of Additional Experimental Formulations Relative to the Micronized Crystalline Tablet in Healthy Subjects
Brief Title: Relative Bioavailability Study With BMS-955176
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 206740; 2013-004896-10 (EudraCT Number); AI468-034 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — BMS-955176

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Cohort 1 Arm ABDC: BMS-955176 (Treatment A, B, D and C) (Experimental): BMS-955176 single dose by mouth as specified
  Interventions: Drug: BMS-955176
- Cohort 1 Arm BCDA: BMS-955176 (Treatment B, C, D and A) (Experimental): BMS-955176 single dose by mouth as specified
  Interventions: Drug: BMS-955176
- Cohort 1 Arm DABC: BMS-955176 (Treatment D, A, B and C) (Experimental): BMS-955176 single dose by mouth as specified
  Interventions: Drug: BMS-955176
- Cohort 1 Arm CDAB: BMS-955176 (Treatment C, D, A and B) (Experimental): BMS-955176 single dose by mouth as specified
  Interventions: Drug: BMS-955176
- Cohort 2 Arm EFGH: BMS-955176 (Treatment E, F, G and H) (Experimental): BMS-955176 single dose by mouth as specified
  Interventions: Drug: BMS-955176
- Cohort 2 Arm FGHE: BMS-955176 (Treatment F, G, H and E) (Experimental): BMS-955176 single dose by mouth as specified
  Interventions: Drug: BMS-955176
- Cohort 2 Arm HEFG: BMS-955176 (Treatment H, E, F and G) (Experimental): BMS-955176 single dose by mouth as specified
  Interventions: Drug: BMS-955176
- Cohort 2 Arm GHEF: BMS-955176 (Treatment G, H, E and F) (Experimental): BMS-955176 single dose by mouth as specified
  Interventions: Drug: BMS-955176

INTERVENTIONS:
Drug: BMS-955176 — BMS-955176

SUMMARY:
The purpose of this study is to select the best dose level (amount of drug given) and best formulation of the study drug (BMS-955176) to develop further.

DETAILED DESCRIPTION:
Primary Purpose: Other: This study will assess the bioavailability of BMS-955176 from a micronized crystalline (MC) tablet relative to a spray-dried dispersion (SDD) suspension. Assessment of additional experimental formulations relative to the micronized crystalline tablet will also be performed

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examinations, vital sign measurements, 12-lead electrocardiogram (ECG) measurements and clinical laboratory test results
* Body mass index (BMI) of 18.0 to 32.0 kg/m2, inclusive. BMI = Weight (kg) / [height (m)]2
* Men and women, ages 18 to 50 years, inclusive
* Women must not be of childbearing potential, must not be breastfeeding

Exclusion Criteria:

* Any significant acute or chronic medical illness
* History of cardiac disease or clinically significant cardiac arrhythmias
* Current or recent (within 3 months of study drug administration) gastrointestinal disease
* Any major surgery within 4 weeks of study drug administration
* Any gastrointestinal surgery (including cholecystectomy) that could impact upon the absorption of study drug

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2014-03-25 (Actual); Primary Completion 2014-07-07 (Actual); Study Completion 2014-07-07 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-955176 | Days 1-4 of Periods 1, 2, 3 and 4
Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of BMS-955176 | Days 1-4 of Periods 1, 2, 3 and 4
Area under the plasma concentration-time curve from time zero to 72 hours post-dose [AUC(0-72)] of BMS-955176 | Days 1-4 of Periods 1, 2, 3 and 4

SECONDARY OUTCOMES:
Time of maximum observed plasma concentration (Tmax) of BMS-955176 | Days 1-4 of Periods 1, 2, 3 and 4
Terminal plasma half-life (T-HALF) of BMS-955176 | Days 1-4 of Periods 1, 2, 3 and 4
Apparent total body clearance (CLT/F) of BMS-955176 | Days 1-4 of Periods 1, 2, 3 and 4
Safety and tolerability based on incidence of adverse events (AEs), serious AEs, AEs leading to discontinuation and deaths, marked abnormalities in clinical laboratory tests, vital sign measurements, ECGs and physical examinations | Up to Period 4/Day 4 (discharge)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Nottingham, United Kingdom